CLINICAL TRIAL: NCT02610816
Title: Eosinophilic Esophagitis (EoE) Intervention Trial-Randomized 1 Food Elimination vs. 4 Food Elimination Diet Followed by Swallowed Glucocorticoids
Brief Title: Eosinophilic Esophagitis Intervention Trial-1 Food vs. 4 Food Elimination Diet Followed by Swallowed Glucocorticoids
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015-2187
Record Dates: First submitted 2015-10-12; First posted 2015-11-20 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Eosinophilic Esophagitis; Eosinophilic Gastrointestinal Disorders (EGIDs)
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1FED (Active Comparator): 1-food elimination diet: Participants eliminate milk from the diet in Phase 1
  Interventions: Other: 1 Food Elimination Diet
- 4FED (Active Comparator): 4-food elimination diet: Participants eliminate milk, egg, wheat, soy from the diet in Phase 1
  Interventions: Other: 4 Food Elimination Diet
- 1FED Non-Responders (4FED) (Other): Participants that fail to respond to 1FED in Phase 1 eliminate milk, egg, wheat, soy from the diet in Phase 2
  Interventions: Other: 4 Food Elimination Diet (post 1FED failure)
- 4FED Non-Responders (SGC) (Other): Participants that fail to respond to 4FED in Phase 1 administer swallowed glucocorticosteroids (Flovent HFA) 800 mcg twice daily in Phase 2
  Interventions: Drug: Fluticasone Propionate, 800 mcg twice daily (post 4FED failure)

INTERVENTIONS:
Other: 1 Food Elimination Diet — Participants eliminate milk from the diet for 12 weeks
  Other Names: 1FED
  Arms: 1FED
Other: 4 Food Elimination Diet — Participants eliminate milk, egg, wheat, soy from the diet for 12 weeks
  Other Names: 4FED
  Arms: 4FED
Other: 4 Food Elimination Diet (post 1FED failure) — Participants that fail to respond to 1FED in phase 1 eliminate milk, egg, wheat, soy from the diet for 12 weeks in Phase 2
  Arms: 1FED Non-Responders (4FED)
Drug: Fluticasone Propionate, 800 mcg twice daily (post 4FED failure) — Participants that fail to respond to 4FED in phase 1 administer swallowed glucocorticosteroids (Flovent HFA) 800 mcg twice daily for 12 weeks in Phase 2
  Arms: 4FED Non-Responders (SGC)

SUMMARY:
The purpose of this interventional study is to test and compare the effectiveness of two elimination diets-the 1-food elimination diet (1FED, milk only) and the 4-food elimination diet (4FED, milk, egg, wheat, and soy) for eosinophilic esophagitis (EoE). The study will also test the effectiveness of swallowed glucocorticoid therapy in some of the study participants for whom diet therapy was not effective.

DETAILED DESCRIPTION:
This study will consist of two phases, plus a screening period. During the screening period, subject eligibility for the study will be determined. During Phase 1, qualified participants will be randomly assigned to one of two elimination diet therapies--the 1FED or the 4FED. Participants will remain on the assigned dietary therapy for 12 weeks. At the end of 12 weeks of therapy, esophageal biopsies from participant's standard of care (i.e. normal, routine care) endoscopy will be evaluated to determine disease status. Participants whose EoE is in remission (i.e. <15 eos/hpf) will be done with the study.

Participants whose EoE is still active (i.e. ≥15 eos/hpf) will continue into Phase 2 of the study. During Phase 2, participants who were on 1FED in Phase 1 will receive 4FED therapy for 12 weeks, and participants who were on 4FED during Phase 1 will receive swallowed glucocorticoid therapy for 12 weeks. At the end of 12 weeks of therapy, esophageal biopsies from participant's standard of care (i.e. normal, routine care) endoscopy will be evaluated to determine disease status.

ELIGIBILITY:
Inclusion Criteria:

* Have diagnosis of EoE (based on consensus criteria)
* Are aged 6 to 17 years
* Have histologically confirmed active disease >15 eosinophils/hpf in either distal or proximal esophagus within 12 weeks of screening visit
* Proton Pump Inhibitor (PPI) confirmation
* Symptomatic (have experienced symptoms within the last month prior to enrollment)
* Has a negative urine pregnancy test at screening if of childbearing potential. Females of childbearing potential must have a negative urine pregnancy test (β-hCG) prior to enrollment into the study (i.e., at screening). Subsequently, these participants must agree to use adequate birth control measures (e.g., condom, oral/injectable/subcutaneous contraceptives, intrauterine device, or sexual abstinence) during the study and for at least one month after the last dose of study drug which will be documented in the source documents.

Exclusion Criteria:

* Have been treated with topical swallowed steroids within the last 2 months or systemic steroids within the past 3 months
* Have eosinophilia in segments of the GI tract other than the esophagus
* Have been diagnosed with a GI malabsorption disorder (i.e., Inflammatory bowel disease, Crohn's disease) or Celiac disease
* Are currently on dietary therapy avoiding milk
* Have concurrent H pylori gastritis or parasitic infection
* Are unable to obtain esophagogastroduodenoscopy with esophageal biopsies at Cincinnati Children's Hospital Medical Center (CCHMC) or other participating institution within 4 weeks of study completion
* Have previously failed (in a clinical trial setting) dietary therapy with one of these regimens or topical steroid treatment with fluticasone at a total dose of 1760 mcg per day.
* Have definitely responded (in a clinical trial setting) to either dietary therapy avoiding these antigens or to swallowed fluticasone at a total dose of 1760 mcg per day
* Are concurrently receiving any of the prohibited medications listed in Table 2
* On immunotherapy for pollen (if not on maintenance therapy) or immunoglobulin E (IgE)-mediated food allergy.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc E Rothenberg, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
The raw anonymized data tables, data dictionaries, and study documentation will be provided to outside investigators upon request, with the proviso that it may not be linked with external datasets so as to minimize the risk of re-identification. When the resources and the associated research findings have been published, data will be made available for research purposes to qualified individuals within the scientific community. Consortium participants will retain rights to any subject inventions generated.
Supporting Information: Study Protocol, SAP
Time Frame: After the associated research findings have been published, data will be made available for research purposes
Access Criteria: Data will be provided in a form suitable for a variety of databases. Data will be provided to qualified individuals within the scientific community, according to federal guidelines.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from eosinophilic esophagitis (EoE) specialty clinics (10 sites) in the USA between November 2015 and February 2018.
Pre-assignment Details: 67 participants screened, 4 excluded (2 did not meet inclusion criteria, 2 met exclusion criteria), and 63 randomized
Groups:
- 1FED: 1-food elimination diet: participants eliminate milk from the diet for 12 weeks
- 4FED: 4-food elimination diet: participants eliminate milk, egg, wheat, soy from the diet for 12 weeks
- 1FED Non-responders (4FED): Participants that fail to respond to 1FED in phase 1 eliminate milk, egg, wheat, soy from the diet for 12 weeks in phase 2
- 4FED Non-responders (SGC): Participants that fail to respond to 4FED in phase 1 administer swallowed glucocorticosteroids (Flovent HFA) 800 mcg twice daily for 12 weeks in phase 2
Period: Phase 1
Arm/Group | 1FED | 4FED | 1FED Non-responders (4FED) | 4FED Non-responders (SGC)
Started | 38 | 25 | 0 | 0
Completed | 34 | 17 | 0 | 0
Not Completed | 4 | 8 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 6 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Period: Phase 2
Arm/Group | 1FED | 4FED | 1FED Non-responders (4FED) | 4FED Non-responders (SGC)
Started | 0 | 0 | 19 | 10
Completed | 0 | 0 | 8 | 4
Not Completed | 0 | 0 | 11 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 9 | 3
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1FED | 4FED | Total
Number analyzed (Participants) | 38 | 25 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.3 (3.1) | 12.1 (3.7) | 12.2 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 26 | 16 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 33 | 21 | 54
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 33 | 22 | 55
  Black or African American | 4 | 1 | 5
  Other | 1 | 2 | 3
Atopy [Count of Participants; unit: Participants]
  Atopic | 34 | 19 | 53
  Not Atopic | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pediatric EoE Symptom Score Version 2.0 (PEESS V2.0) at 12 Weeks
Description: The PEESS V2.0 questionnaire captures EoE-specific symptoms (dysphagia, gastro-esophageal reflux disease (GERD), nausea/vomiting, and pain) as reported by children with EoE (8-18 years of age) and their parents (for children 2-18 years of age). The range for PEESS v2.0 scores is 0 to 100, with a higher score being indicative of more frequent and/or severe symptoms. Scores were obtained at baseline and 12 weeks. Change in score is defined as total score at 12 weeks minus total score at baseline. The parent-proxy PEESS total score change from pre-treatment to post-treatment is the primary efficacy endpoint. 1FED vs 4FED changes are compared. A reduction in score (negative change) is indicative of a reduction in symptoms.
Time Frame: Baseline and 12 weeks
Population: We performed intent to treat analysis including participants who had at least one clinical observation post randomization.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1FED | 4FED
Number analyzed (Participants) | 33 | 16
units on a scale | -14.3 (17.1) | -21.6 (17.3)
Statistical Analysis 1: Comparison: 1FED vs 4FED; The primary treatment comparison was to compare change in PEESS V2.0 scores of 1FED versus 4FED. The primary null hypothesis was 4FED would be no more effective than 1FED. This was designed as a superiority trial; Test type: Superiority; p = 0.04, Mixed Models Analysis — P-values are not adjusted for multiplicity, since a single primary endpoint is analyzed; No adjustment of degrees of freedom is needed

2. Primary Outcome: Within-group Comparisons (Baseline v. Week 12) of PEESS V2.0 Scores
Description: The PEESS V2.0 questionnaire captures EoE-specific symptoms. The range for PEESS v2.0 scores is 0 to 100, with a higher score being indicative of more frequent and/or severe symptoms. Baseline vs Week 12 scores are compared within each treatment group (1FED and 4FED).
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1FED | 4FED
Number analyzed (Participants) | 38 | 24
units on a scale
  Baseline - Total Score | 38.1 (14.2) | 42.9 (16.0)
  Week 12 - Total Score: number analyzed (Participants) | 33 | 17
  Week 12 - Total Score | 23.5 (18.3) | 16.0 (13.0)
Statistical Analysis 1: Comparison: 1FED; Test type: Superiority; p < 0.0001, Mixed Models Analysis — This is a calculated p-value. The threshold for statistical significance is p <0.05
Statistical Analysis 2: Comparison: 4FED; Test type: Superiority; p < 0.0001, Mixed Models Analysis — This is a calculated p-value. The threshold for statistical significance is p <0.05

3. Secondary Outcome: Percent of Participants in Histologic Remission (<15 Eosinophils Per High Power Field) at 12 Weeks
Description: Percent of participants in remission in 1FED and 4FED groups. Remission is defined as clinical esophageal peak eosinophil count < 15 eosinophils per high power field (eos/hpf). Complete remission is defined as ≤ 1 peak eos/hpf and partial remission as 2 - 14 peak eos/hpf.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 1FED | 4FED
Number analyzed (Participants) | 34 | 17
percentage of participants
  Complete remission (≤ 1 eos/hpf) | 20.6 | 17.6
  Partial remission (2 - 14 eos/hpf) | 23.5 | 23.5
  Remission (< 15 eos/hpf) | 44.1 | 41.2
Statistical Analysis 1: Comparison: 1FED vs 4FED; Test type: Superiority; p = 1.0, Fisher Exact

4. Secondary Outcome: Percent of Participants on Swallowed Glucocorticoids (SGC) in Histologic Remission (<15 Eos/Hpf) at 12 Weeks in Phase 2
Description: Percent of 4FED non-responders on SGC in Phase 2 in histologic remission. Remission is defined as esophageal peak eosinophil count < 15 eosinophils per high power field (eos/hpf). Complete remission is defined as ≤ 1 peak eos/hpf and partial remission as 2 - 14 peak eos/hpf.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 4FED Non-responders (SGC)
Number analyzed (Participants) | 4
percentage of participants
  Complete remission (≤ 1 eos/hpf) | 25.0
  Partial remission (2 - 14 eos/hpf) | 25.0
  Remission (< 15 eos/hpf) | 50.0

5. Secondary Outcome: Percent of 1FED Non-responders on 4FED in Histologic Remission (<15 Eos/Hpf) at 12 Weeks in Phase 2
Description: Percent of 1FED non-responders on 4FED in histologic remission in phase 2. Remission is defined as esophageal peak eosinophil count < 15 eosinophils per high powered field. Complete remission is defined as ≤ 1 peak eos/hpf and partial remission as 2 - 14 peak eos/hpf.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 1FED Non-responders (4FED)
Number analyzed (Participants) | 8
percentage of participants
  Complete remission (≤ 1 eos/hpf) | 0
  Partial remission (2 - 14 eos/hpf) | 12.5
  Remission (< 15 eos/hpf) | 12.5

6. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Inventory Version 3.0 EoE Module (PedsQL 3.0 EoE) at 12 Weeks
Description: The PedsQL 3.0 EoE measures symptoms and problems related to treatment, worry, communication, food/eating, and feelings. The range for PedsQL 3.0 EoE scores is 0 to 100, with a higher score indicating better quality of life. Scores were obtained at baseline and 12 weeks. Change in score is defined as the PedsQL 3.0 EoE total score at 12 weeks minus total score at baseline. 1FED vs 4FED changes are compared. An increase in score (positive change) is indicative of improved quality of life.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1FED | 4FED
Number analyzed (Participants) | 38 | 25
units on a scale
  Baseline - Total Score | 71.3 (13.0) | 67.5 (13.6)
  Change from Baseline to Week 12: number analyzed (Participants) | 31 | 16
  Change from Baseline to Week 12 | 9.7 (11.3) | 9.8 (14.1)
Statistical Analysis 1: Comparison: 1FED vs 4FED; Test type: Superiority; p = 0.93, Mixed Models Analysis

7. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Inventory Version 4.0 (PedsQL 4.0) Generic Core Scales at 12 Weeks
Description: The PedsQL 4.0 measures physical and psychosocial function. The range for PedsQL 4.0 scores is 0 to 100, with a higher score indicating better quality of life. Scores were obtained at baseline and 12 weeks. Change in score is defined as the PedsQL 4.0 total score at 12 weeks minus total score at baseline. 1FED vs 4FED changes are compared. An increase in score (positive change) is indicative of improved quality of life.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1FED | 4FED
Number analyzed (Participants) | 38 | 24
units on a scale
  Baseline - Total Score | 80.3 (10.8) | 79.9 (14.5)
  Change from Baseline to Week 12: number analyzed (Participants) | 33 | 16
  Change from Baseline to Week 12 | 3.7 (9.9) | 5.3 (16.4)
Statistical Analysis 1: Comparison: 1FED vs 4FED; Test type: Superiority; p = 0.74, Mixed Models Analysis

8. Secondary Outcome: Change From Baseline in Endoscopic Reference Score at 12 Weeks
Description: The EoE Endoscopic Reference Score (EREFS) measures features of EoE including esophageal edema, rings, exudate, furrows, and strictures. The instrument grades edema and furrows as absent (0) or present (1); rings as absent (0), mild (1, subtle circumferential ridges), moderate (2, distinct rings) and severe (3, rings that impair passage of a standard adult diagnostic endoscope); exudates as absent (0), mild (1, less than 10% of the esophageal surface area) or severe (2, greater or equal to 10% of the esophageal surface area); and strictures as absent (0) or present (1) with an estimation of the minimal luminal diameter. Higher scores indicate more severe disease (range 0 - 9). Scores were obtained at baseline and 12 weeks. Change in score is defined as the EREFS total score at 12 weeks minus total score at baseline. 1FED vs 4FED changes are compared. A reduction in score (negative change) is indicative of a reduction in esophageal abnormalities.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1FED | 4FED
Number analyzed (Participants) | 22 | 12
units on a scale
  Baseline - Total Score | 2.5 (1.3) | 3.3 (1.8)
  Change from Baseline to Week 12: number analyzed (Participants) | 17 | 12
  Change from Baseline to Week 12 | -0.7 (2.2) | -1.3 (2.2)
Statistical Analysis 1: Comparison: 1FED vs 4FED; Test type: Superiority; p = 0.36, Mixed Models Analysis

9. Secondary Outcome: Percent of Participants With Positive and Negative Milk Skin Prick Tests Responding to 1FED
Description: Reactions to skin prick test (SPT) to milk is positive if the wheal size of the milk test is at least 3 mm larger than the wheal size of the negative control. Treatment response is defined as clinical histologic remission (<15 eos/hpf).
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 1FED
Number analyzed (Participants) | 28
percentage of participants
  Percent of total with positive milk SPT | 11
  Percent of total with negative milk SPT | 89
  Percent with positive SPT responding to 1FED | 33
  Percent with negative SPT responding to 1FED | 48

ADVERSE EVENTS:
Time Frame: Adverse events were collected from informed consent/assent to 30 days after the cessation of the study agent (2 years, 2 months).
Groups:
- 1FED: 1-food elimination diet (Phase 1)
- 4FED: 4-food elimination diet (Phase 1)
- 1FED Non-responders (4FED): 4-food elimination diet (Phase 2)
- 4FED Non-responders (SGC): Swallowed glucocorticosteroids (Flovent HFA) (Phase 2)
Arm/Group | 1FED | 4FED | 1FED Non-responders (4FED) | 4FED Non-responders (SGC)
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/25 | 0/19 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/38 | 1/25 | 0/19 | 0/10
Other Adverse Events (participants affected / at risk) | 5/38 | 8/25 | 6/19 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1FED (N=38) | 4FED (N=25) | 1FED Non-responders (4FED) (N=19) | 4FED Non-responders (SGC) (N=10)
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1FED (N=38) | 4FED (N=25) | 1FED Non-responders (4FED) (N=19) | 4FED Non-responders (SGC) (N=10)
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Otitis Media (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT02610816/Prot_000.pdf
  • Statistical Analysis Plan (2015-03-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT02610816/SAP_001.pdf